CLINICAL TRIAL: NCT04996758
Title: An Open-Label, Phase Ⅱ Study of Toripalimab and Anlotinib Combination Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma After Failure of at Least One Line of Platinum-Based Chemotherapy (TORAL)
Brief Title: Toripalimab and Anlotinib Combination Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma After Failure of at Least One Line of Platinum-Based Chemotherapy (TORAL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-055
Record Dates: First submitted 2021-08-05; First posted 2021-08-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent or Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — toripalimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab and Anlotinib Combination Treatment (Experimental): Patients receive toripalimab at a dose of 240 mg on day 1 and anlotinib at a dose of 12 mg before breakfast for once-daily on days 1-14. Treatment cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: Toripalimab and Anlotinib

INTERVENTIONS:
Drug: Toripalimab and Anlotinib — Toripalimab 240 mg iv.drip d1; Anlotinib 12mg po qd d1-14.

SUMMARY:
This phase 2 trial studies toripalimab and anlotinib combination treatment in patients with recurrent or metastatic nasopharyngeal carcinoma after failure of at least one line of platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed undifferentiated non-keratinizing carcinoma
* Patients suffered failure of at least one line of platinum-based chemotherapy. The definition of treatment failure: progression during or after chemotherapy for recurrence/metastasis; progression after concurrent chemoradiotherapy within 6 months. Withdrawal of treatment due to drug intolerances is excluded ;
* Without other malignancy;
* Male or female, 18-70 years;
* Eastern Cooperative Oncology Group (ECOG) of 0-2;
* Life expectancy ≥ 3 months;
* Women of childbearing age must obtain the negative result of a pregnancy test (serum or urine) , and they were willing to use reliable methods of contraception during the trial;
* At least one evaluable lesion；
* Laboratory tests meet the following standards:

Blood routine: White blood cell count (WBC) ≥3.0×10 9 /L, neutrophil count (ANC) ≥1.5×10 9 /L, platelet count (PLT) ≥75×10 9 /L, hemoglobin (HGB) 90 g/L or higher; Liver function: total bilirubin ≤1.5 times the upper limit of normal (ULN); glutamic-oxalacetic transaminase (AST) and alanine transaminase (ALT) ≤2.5 times ULN, AST and ALT ≤2.5 times ULN for the patients with liver metastases; Alkaline phosphatase ≤5 times ULN; Renal function: Serum creatinine (Cr) ≤1.5 times ULN; Creatinine clearance ≥60mL/min; Urine routine: urine protein <2+ ;baseline urine protein ≥2+ and 24 hours urine protein < 1g ; Coagulation: International normalized ratio (INR) and activated partial thrombin time (APTT) ≤1.5 times ULN; Albumin ≥28g/L Thyroid stimulating hormone (TSH)≤1 times ULN (free triiodothyrosine [FT3] or free thyroxine [FT4] ≤1 times ULN can be included)

* No serious cardiopulmonary dysfunction;
* The informed consent has been signed.
* Ability to comply with test requirements

Exclusion Criteria:

* A known allergy to any of the drugs in the study;
* Pregnant or breastfeeding women;
* Participated in clinical trials of other drugs within 4 weeks prior to study initiation;
* Previous treatment with bevacizumab or VEGFR-family small molecule tyrosine kinase inhibitors (e.g., famitinib, sorafenib, Sunitinib, regofinib, Apatinib, Anlotinib, fuquinitinib) ;
* Recurrent nasopharyngeal lesions after radiotherapy and who received secondary radiotherapy;
* Palliative radiotherapy for symptom control within 28 days before enrollment;
* Immunosuppressive treatment with immunosuppressive agent, systemic or absorbable topical hormone therapy ( prednisone or other therapeutic hormone at the dose greater than 10mg/ day) within 2 weeks before enrollment;
* Active autoimmune diseases, with the necessity of systemic treatment (hormone replacement therapy is not considered as a systemic treatment, such as type 1 diabetes) over the past two years; autoimmune diseases that did not require systemic treatment in the past two years;
* A history of immunodeficiency, including acquired/congenital immunodeficiency disorders, a history of organ transplantation;
* Vaccinated with live vaccine (inactivated virus vaccine for seasonal influenza is allowed) within 4 weeks before enrollment;
* Invasion of important vessels (e.g. surrounding internal carotid artery/vein) on MRI; tumor with a high risk of affecting vital blood vessels during treatment and causing fatal hemorrhage, which is determined by investigators;
* A history of severe bleeding and any bleeding event with a severity rating of 3 or higher in the NCI CTCAE within 4 weeks prior to screening;
* Abnormal coagulation (INR > 2.0, PT > 16s) and bleeding tendency (the INR must be within the normal range without anticoagulants during14 days prior to signing the informed consent); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogests; low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (up to 100 mg daily) for preventive purposes, provided that the international normalized ratio of prothrombin time (INR) is ≤ 1.5;
* Unstable angina and/or congestive heart failure or vascular disease with the need of hospital treatment; other cardiac damage that may affect the drug safety;
* Patients with hypertension that is not well controlled with antihypertensive medication (systolic > 140mmHg, diastolic > 90 mmHg); patients is taking a combination of two or more antihypertensive drugs; Cardiovascular disease with clinical significance， such as cerebrovascular accident (≤ 6 months before randomization), myocardial infarction (≤ 6 months before randomization), unstable angina, congestive heart failure of NYHA grade II or higher, or severe arrhythmias that cannot be controlled with drugs or have a potential impact on experimental treatments;
* Patients with esophageal and gastric varices, active ulcers, intestinal perforation or intestinal obstruction within 6 months before enrollment;
* A history of abdominal fistula, digestive tract perforation, intra-abdominal abscess or acute gastrointestinal bleeding within 6 months before enrollment;
* Multiple factors affecting oral administration and absorption of drugs (e.g., inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction);
* Overoperation/venous thromboembolism events, NCI CTCAE grade 3 or higher venous thromboembolism within 6 months before enrollment, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except for those venous thrombosis caused by venous catheterization due to previous chemotherapy and determined to be cured by the researchers ), pulmonary embolism, etc.;
* Patients with past and present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe impairment of lung function;
* Exacerbation of chronic obstructive pulmonary disease (COPD) or other respiratory disease requiring hospitalization within 28 days before enrollment;
* Active pulmonary infection and/or acute bacterial or fungal infection requiring intravenous antibiotic treatment within 28 days;
* Dominant jaundice due to abnormal liver function within 7 days;
* Renal insufficiency: routine urinalproteinuria > 2+ and confirmed 24 h urinary protein quantification > 1.0g;
* Minor surgical operations (including catheterization, excluding central venous catheterization via peripheral venipuncture) within 2 days before enrollment;
* Major surgery within 28 days before enrollment;
* A potent CYP3A4 inhibitor within one week prior to enrollment, or a potent CYP3A4 inducer within two weeks prior to study participation
* Long-term unhealed wounds or incomplete fractures;
* Symptomatic central nervous system metastases (e.g. brain edema, need for hormonal intervention, or brain metastases)
* The presence of serious or uncontrolled infections;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Objective Response rate | 2 years
  Objective Response rate will be determined on the basis of investigator assessments

SECONDARY OUTCOMES:
Disease Control rate | 2 years
  the proportion of patients who had a best response rating of complete response, partial response, or stable disease will be determined on the basis of investigator assessments
Progression Free Survival | 5 years
  The time from the start of treatment to the progression of the tumor or death (due to any cause).
Overall Survival | 5 years
  The time from the start of treatment to time of death (due to any cause).
Complete Response rate | 2 years
  Complete Response rate will be determined on the basis of investigator assessments
Partial Response rate | 2 years
  Partial Response rate will be determined on the basis of investigator assessments
Duration of Response | 5 years
  The time from the first assessment of complete remission or partial remission to progressive disease or death (due to any cause).
Percentage of Participants With Adverse Events | 5 years
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, Principal Investigator — Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, China

REFERENCES:
- [Derived] Zhang Y, Zou Q, Zhao B, Su N, Li Z, Wang X, Liu P, Tian X, Fang X, Cai J, Li L, Liu Y, Xia Y, Cai Q. Toripalimab plus anlotinib in patients with recurrent or metastatic nasopharyngeal carcinoma: A multicenter, single-arm phase 2 trial (TORAL). Cell Rep Med. 2024 Dec 17;5(12):101833. doi: 10.1016/j.xcrm.2024.101833. Epub 2024 Nov 29. PMID 39615484